CLINICAL TRIAL: NCT00267904
Title: Reference Values for Plasma Catechols
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 060047; 06-N-0047
Record Dates: First submitted 2005-12-21; First posted 2005-12-21 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers; Normal Physiology
Keywords: Adrenaline; Normal Physiology; Catecholamines; Catechols; Sympathetic Nervous System; Healthy Volunteer; HV
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy Volunteer for Banana (Experimental): Ingestion of a single banana
  Interventions: Other: Banana
- Healthy Volunteer for Coffee (Experimental): Ingestion of caffeinated coffee on one day and decaffeinated coffee on another day
  Interventions: Other: Coffee
- Healthy Volunteer for Olive (Experimental): Ingestion of olives
  Interventions: Other: Olives
- Healthy Volunteer for Quality Control Plasma (No Intervention): Arm venous blood is drawn via an indwelling i.v. catheter from HVs to obtain quality control plasma
- Healthy Volunteer for Temp. Manip. (Experimental): Manipulation of temperature at skin of the back
  Interventions: Other: Temp. manip.

INTERVENTIONS:
Other: Coffee — Caffeinated coffee and decaffeinated coffee ingestion
  Arms: Healthy Volunteer for Coffee
Other: Banana — Banana ingestion
  Arms: Healthy Volunteer for Banana
Other: Olives — Olives ingestion
  Arms: Healthy Volunteer for Olive
Other: Temp. manip. — Manipulate temperature at skin of the back
  Arms: Healthy Volunteer for Temp. Manip.

SUMMARY:
Objectives: Plasma levels of catechols have distinct meanings in terms of indicating functions of endogenous catecholamine systems. This Protocol is designed to enable ongoing quality assurance of diagnostic and research assays of catechols and their metabolites and to identify possible influences of demographic and anthropometric factors, dietary constituents, and conditions of sampling on reference values.

Study Populations: The study population is healthy volunteers and people who are obese or have untreated hypertension.

Design: Arm venous blood is drawn via an indwelling i.v. catheter from healthy volunteers across demographic and anthropometric spectra (age, gender, skin color, ethnicity, body mass, adiposity), to obtain quality control plasma and establish reference values for plasma levels of catechols and their metabolites. Non-invasive physiological measures are obtained concurrently. Levels of catechols and their metabolites are related to results of common clinical pathology tests. Subgroups of subjects are tested more than once, to assess dietary influences (cereal with milk, coffee) and conditions of sampling (temperature at the skin).

Outcome Measures: The main non-experimental outcome is an ongoing pool of quality control plasma. The main experimental outcome measures are plasma concentrations of catechols and their metabolites, non-invasive physiological measures, and results of common clinical pathology tests. Subject groups are compared with respect to the above demographic and anthropometric factors. Effects of the experimental manipulations are assessed within subjects

DETAILED DESCRIPTION:
Objective: Plasma levels of catechols have distinct meanings in terms of indicating functions of endogenous catecholamine systems. This protocol is designed to enable ongoing quality assurance of diagnostic and research assays of catechols and their metabolites and to identify possible influences of dietary constituents and conditions of sampling.

Study Population:The study population is Healthy Volunteers (HVs).

Design: Arm venous blood is drawn via an indwelling i.v. catheter from HVs to obtain quality control plasma. Levels of catechols and their metabolites are related to dietary influences (e.g., coffee, olives, banana) and conditions of sampling (temperature at the skin) by repeated measurements in the same subjects over time.

Outcome Measures: The main non-experimental outcome is an ongoing pool of quality control plasma. The main experimental outcome measures are plasma concentrations of catechols and their metabolites and physiological measures, and results of common clinical pathology tests. Effects of the experimental manipulations are assessed within subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

The subjects are healthy volunteers 18 years or older who are not pregnant or lactating.

EXCLUSION CRITERIA:

<TAB>

Minors younger than 18 years old are excluded.

A candidate subject is excluded if, in the judgment of the Principal Investigator, Protocol participation would place the subject at substantially increased acute medical risk. A candidate subject is excluded if, in the opinion of the Principal Investigator, the medical risk outweighs the potential scientific benefit.

A candidate subject is excluded if there is a disqualifying condition. Examples of disqualifying conditions are hepatic failure, a history of tachyarrhythmias or heart block, symptomatic congestive heart failure, severe anemia, psychosis, refractory ventricular arrhythmias, symptomatic coronary heart disease, diabetes mellitus, or hyperthyroidism. Abnormal screening results may exclude further participation, at the discretion of the Principal Investigator.

Subjects will be excluded from further participation and referred for medical management, if the systolic blood pressure during supine rest is greater than or equal to 160 mm Hg or diastolic blood pressure greater than or equal to 105 mm Hg.

Alcohol use disorder.

A candidate subject is excluded if clinical considerations require that the patient continue treatment with a drug likely to interfere with the scientific results. Examples are acetaminophen, angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, adrenoceptor agonists or antagonists, anticoagulants, anticonvulsants, antipsychotics, calcium channel blockers, hypoglycemic agents, digoxin, dopaminergic drugs, monoamine oxidase inhibitors, oral contraceptives, sedatives, steroids, and tricyclic antidepressants. Patients are not to discontinue any medications, just to participate in this study.

Subjects in whom we feel it would be difficult to insert a catheter into a vein may be excluded.

Pregnant or lactating women are excluded. To exclude pregnancy, women with child bearing potential have blood testing for pregnancy, with negative results obtained within 1 day of each day of testing.

Candidate subjects who admit to a history of alcohol addiction and alcohol use disorder are excluded from the study as a whole, but is especially important in the portion of the study involving ingesting red wine.

Candidate subjects who drink alcohol every day are excluded from the portion of the study involving ingesting red wine.

People with a history of sulfite allergy are excluded from the portion of the study involving ingestion of red wine.

Subjects must be at least 21 years old in order to participate in the portion of the study involving ingestion of red wine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-03-08 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Pool of quality control plasma | One time (over 1-4 outpatient visits)
  The main non-experimental outcome is an ongoing pool of quality control plasma.
Plasma concentrations of catechols and their metabolites and physiological measure | One time (over 1-4 outpatient visits)
  The main experimental outcome measures are plasma concentrations of catechols and their metabolites and physiological measures, and results of common clinical pathology tests. Effects of the experimental manipulations are assessed within subjects.

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldstein, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstein DS, Lenders JW, Kaler SG, Eisenhofer G. Catecholamine phenotyping: clues to the diagnosis, treatment, and pathophysiology of neurogenetic disorders. J Neurochem. 1996 Nov;67(5):1781-90. doi: 10.1046/j.1471-4159.1996.67051781.x. PMID 8863481
- [Background] Eisenhofer G, Goldstein DS, Stull R, Keiser HR, Sunderland T, Murphy DL, Kopin IJ. Simultaneous liquid-chromatographic determination of 3,4-dihydroxyphenylglycol, catecholamines, and 3,4-dihydroxyphenylalanine in plasma, and their responses to inhibition of monoamine oxidase. Clin Chem. 1986 Nov;32(11):2030-3. PMID 3096593
- [Background] Holmes C, Eisenhofer G, Goldstein DS. Improved assay for plasma dihydroxyphenylacetic acid and other catechols using high-performance liquid chromatography with electrochemical detection. J Chromatogr B Biomed Appl. 1994 Mar 4;653(2):131-8. doi: 10.1016/0378-4347(93)e0430-x. PMID 8205240
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2006-N-0047.html